CLINICAL TRIAL: NCT06622460
Title: Experimental Evaluation of the Virtual Eggs Test on Healthy Participants
Brief Title: VET Evaluation: Healthy
Acronym: VET_Healthy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Unknown)
Responsible Party: Principal Investigator, Francesca Cecchi, MD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VirtualEggTest_Healthy
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Hand Control Group (HHC Group) (Experimental): The Healthy Hand Control Group (HHC Group) consists of participants without motor impairments, selected to establish baseline data for hand dexterity and grip strength using the Virtual Eggs Test (VET).
  Interventions: Other: Hand Dexterity Assessment

INTERVENTIONS:
Other: Hand Dexterity Assessment — to evaluate the reliability and sensitivity of the VET in healthy. Their performance helps define normal thresholds and behaviors in grip force modulation and manual dexterity.

SUMMARY:
The study involving healthy participants aims to validate the Virtual Eggs Test (VET) as a tool for measuring hand dexterity and grip force control. This part of the study focuses on determining the test's reliability and validity in a population without motor impairments. Healthy participants will perform the VET using both their dominant and non-dominant hands across two sessions. The purpose is to establish baseline performance metrics for comparison with stroke patients and to assess the test's usability in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years.
* No motor deficits.
* Adequate cognitive and language abilities to understand the experiment and follow instructions.
* Signed informed consent.

Exclusion Criteria:

* Significant visual or oculomotor impairments.
* Comorbidities or disabilities that may interfere with the study, such as multiple sclerosis, Parkinson's disease, or muscle tone disorders.
* Cardiopulmonary or circulatory pathologies.
* Pregnancy or breastfeeding.
* Psychiatric comorbidities.
* Difficulty understanding the Italian language.
* Lack of cooperation.
* Consumption of alcohol or diuretics before the test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Threshold from the Virtual Eggs Test (VET) | First Session (Test)
  This refers to the grip strength threshold required to avoid breaking fragile objects during the test. The VET measures the participant's ability to regulate grip strength and dexterity, with the threshold ranging from 1 to 20. Lower numbers indicate that less force is needed to break the object, reflecting greater control over fine motor skills
Threshold from the Virtual Eggs Test (VET) | Second Session (Re-Test)
  This refers to the grip strength threshold required to avoid breaking fragile objects during the test. The VET measures the participant's ability to regulate grip strength and dexterity, with the threshold ranging from 1 to 20. Lower numbers indicate that less force is needed to break the object, reflecting greater control over fine motor skills

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi ONLUS, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No